CLINICAL TRIAL: NCT06337929
Title: Effects of Capoeira Training on Physical Performance and Psychological Aspects Performance of Adults: a Randomized Controlled Clinical Trial
Brief Title: Effects of Capoeira on the Physical and Psychological Performance of Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do vale do São Francisco (Other)
Responsible Party: Principal Investigator, Sérgio Rodrigues Moreira, Professor (PhD), Universidade Federal do vale do São Francisco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Ethics Approval: n. 6.683.936
Record Dates: First submitted 2024-03-15; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Training; Mental Health; Physical Fitness
Keywords: Combat sports; Brazilian martial art; Physical fitness
MeSH Terms: conditions — Psychological Well-Being | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAPOEIRA GROUP (Experimental): The training program will be conducted over 12 weeks with two weekly sessions. Each session will last 60 minutes and will be divided into three parts: 1) initial part: execution of stretches and low-intensity actions with specific movements of capoeira; 2) main part: realization of the training program the schedule present in Table 1 for the learning of attacks, dodges and acrobatic movements or flourishes and; 3) Final part: in a self-selected way in the capoeira roda, the participant will develop the previously learned movements.
  Interventions: Other: CAPOEIRA TRAINING
- CONTROL GROUP (Active Comparator): The CONTROL GROUP will be conducted over 12 weeks with two weekly sessions. Each session will last 60 minutes and will be divided into three parts: 1) initial part: execution of stretches and low-intensity actions with specific movements of capoeira; 2) main part: continuation with execution of stretches and low-intensity actions with specific movements of capoeira and; 3) Final part: in a self-selected way in the capoeira roda, the participant will develop the previously learned movements.
  Interventions: Other: CONTROL GROUP

INTERVENTIONS:
Other: CAPOEIRA TRAINING — The protocol of the capoeira training program and the movements (blows, dodges and flourishes) will be based on the Capoeira Abadá method.
  Arms: CAPOEIRA GROUP
Other: CONTROL GROUP — The protocol of the control group will be based on an intervention with capoeira movements, however, without important cardiovascular, neuromuscular and metabolic demands, being an activity with stretching movements from positions of the capoeira modality itself.
  Arms: CONTROL GROUP

SUMMARY:
Regular physical activity (PA) promotes benefits for both physical and mental health. Among the numerous PA's with a collective nature that can add to the existing recommendations, combat sports training interventions are viable alternatives since they integrate benefits in different aspects for health. In this way, capoeira can be a strategy for the prescription of exercise, aiming to serve participants collectively and maintaining the adherence of this practitioner to the intervention. However, little is known about this issue. So, the aim of the present study is to verify the effect of 12 weeks of capoeira training on the physical performance and psychological aspects of previously physically inactive adults.

DETAILED DESCRIPTION:
The study will be conducted as a controlled, randomized, two-group parallel and superiority clinical trial with a 1:1 allocation ratio. The sample will be divided into two groups: 1) capoeira training group (n = 76; GCAP) and 2) control group (n = 76; GCONT). Participants aged between 18 and 59 years, classified as irregularly active A by the international physical activity questionnaire, who are not engaged in training programs and are not former athletes, will be eligible. Smokers and patients with respiratory or cardiovascular diseases will be excluded from the sample. Anamnesis and anthropometric evaluation will initially be performed. To evaluate the physical aspects, specific tests will be applied to determine aerobic and anaerobic fitness, strength and power of lower limbs, balance, motor coordination and questionnaires will be applied to verify the psychological aspects, such as emotional intelligence, motivation and quality of life. The descriptive analysis of the outcomes will be reported. The normality of the data will be checked by visual inspection of the Q-Q plot and statistically tested by the Shapiro-Wilk test. Two-way ANOVA for repeated measures will be employed to verify the time*group interaction. The effect size (ES) of the intervention on dependent variables will be calculated and the difference between the ES and its respective 95% confidence interval will be calculated to estimate the magnitude of the response in the intervention. The alpha adopted will be 5% and the software used for data analysis will be Statistical Packages for the Social Sciences 25.0.

ELIGIBILITY:
Inclusion Criteria:

* Classified as "irregularly active A" by the International Physical Activity Questionnaire;
* Do not be engaged and/or have participated in the last two months of any physical training program;
* Do not be former athletes;
* Do not be a smoker or suffering from respiratory or cardiovascular diseases.

Exclusion Criteria:

* Do not have musculoskeletal problems during the program that make it impossible to participate;
* Do not participating in at least 80% of the training sessions during the intervention.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-12-13 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in aerobic fitness (maximal oxygen uptake and anaerobic threshold) at week 12 | Baseline and week 12
  The maximal oxygen uptake and anaerobic threshold are valid indicators for assessing aerobic fitness
Change from baseline in anaerobic fitness (Peak, average and minimum power in the Wingate test) at week 12 | Baseline and week 12
  The Peak, average and minimum power in the Wingate test are valid indicators for assessing anaerobic fitness
Change from baseline in muscle strength (Horizontal Leg Press) at week 12 | Baseline and week 12
  The methods and procedures are valid indicators for assessing muscle strength
Change from baseline in muscle power (Vertical Jump Tests from Squat Jump and Counter Movement Jump) on force platform at week 12 | Baseline and week 12
  The methods and procedures are valid indicators for assessing muscle power
Change from baseline in balance (Center of Pressure) on force platform at week 12 | Baseline and week 12
  The methods and procedures are valid indicators for assessing balance
Change from baseline in motor coordination (Test of Gross Motor Development) at week 12 | Baseline and week 12
  The methods and procedures are valid indicators for assessing motor coordination
Change from baseline in Emotional Intelligence to sport (Likert-type scales with 26 items) at week 12 | Baseline and week 12
  The methods and procedures are valid indicators for assessing Emotional Intelligence with changes 26 (worst) to 130 (better) points
Change from baseline in Motivation for Sport II (Likert-type scales with 18 items) at week 12 | Baseline and week 12
  The methods and procedures are valid indicators for assessing Motivation for Sport with changes 1 (worst) to 7 (better) points
Change from baseline in Quality of life measuring by Questionnaire of Word Health Organization (WHOQOL-bref) at week 12 | Baseline and week 12
  The procedures are valid indicators for assessing Quality of life (26 questions divided into four domains - physical, social, psychological, and environmental) with changes 1 (worst) to 100 (better) points

CONTACTS AND LOCATIONS:
Locations (1):
- UNIVASF, Petrolina, Pernambuco, Brazil